CLINICAL TRIAL: NCT06858059
Title: A Randomized Controlled Trial of the Efficacy of the Lighthouse Parenting Effectiveness Enhancement Programme in Addressing Parenting Difficulties
Brief Title: A Randomized Controlled Trial of the Efficacy of the Lighthouse Parenting Programme in Addressing Parenting Difficulties in China
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-317-03
Record Dates: First submitted 2024-12-17; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-12

CONDITIONS: Parenting Intervention
Keywords: Parenting Intervention
MeSH Terms: interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The test group (Group A) (Experimental): The experimental group will be conducted in the form of assessments, group intervention and individual intervention . All participants will take part in full treatment over a period of five weeks. Each week, participants will engage in one group session lasting approximately 90 minutes and one individual session lasting approximately 60 minutes. A assessment will be conducted at the time of recruitment and following the final individual session.
  Interventions: Other: psychological intervention
- The control group (Group B) (No Intervention): The control group will undergo the same intervention as the test group after the test group completes the intervention and posttest, and will be assessed one additional time for pre-intervention status.

INTERVENTIONS:
Other: psychological intervention — All participants of the lighthouse parenting programme will engage in the full program over a period of five weeks, divided into ten sessions. The 5 group interventions will occur once a week for 1.5 hours. During this time, the psychotherapist will disseminate psychological knowledge and skills pertinent to parenting, after which the group members will engage in practice exercises and discourse. Subsequently, one individual session will be conducted each week for one hour.
  Arms: The test group (Group A)

SUMMARY:
The study will be conducted in three phases: assessments, group intervention and individual intervention. All participants will engage in the full program over a period of five weeks, divided into ten sessions. The 5 group interventions will occur once a week for 1.5 hours. During this time, the psychotherapist will disseminate psychological knowledge and skills pertinent to parenting, after which the group members will engage in practice exercises and discourse. Subsequently, one individual session will be conducted each week for one hour. The test group (Group A) will be assessed once at recruitment and after the last individual session. The control group (Group B) will undergo the same intervention as the test group after the test group completes the intervention and posttest, and will be assessed one additional time for pre-intervention status.

ELIGIBILITY:
Inclusion Criteria:

* Parents with children aged 2-14 years who exhibited parenting that were identified as being problematic (Parenting Stress Indicator PSI ≥ 86 (critical high level)).

Exclusion Criteria:

* Parents in the family with either parent and child who have a serious medical condition (e.g., cancer, heart disease, etc.), an acute psychotic episode, or difficulty engaging in group interventions may be excluded from participation.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-12-13 (Estimated)

PRIMARY OUTCOMES:
Parenting stress | From enrollment to the end of treatment at 5 weeks
  The Parenting Stress Index/Short Form (PSI/SF; Abidin, 1986) is employed to assess parenting stress.

SECONDARY OUTCOMES:
Parental mentalising | From enrollment to the end of treatment at 5 weeks
  The Parental Reflective Functioning Questionnaire (PRFQ; Luyten, Mayes, Nijssens, & Fonagy, 2017) is employed to assess parental mentalizing.
Quality of the parent-child relationship | From enrollment to the end of treatment at 5 weeks
  The quality of the parent-child relationship is evaluated using the Multiperspective Parent-Child Relationship Questionnaire (M-PCR; Müller & Achtergarde, 2018).
parenting efficacy | From enrollment to the end of treatment at 5 weeks
  The Brief Parental Self-Efficacy Scale (Woolgar et al., 2023) is employed to assess parenting efficacy.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Volkert J, Georg A, Hauschild S, Herpertz SC, Neukel C, Byrne G, Taubner S. [Strengthening Attachment Competencies in Parents with Mental Illness: Adaptation and Pilot Testing of the Mentalization-Based Lighthouse Parenting Program]. Prax Kinderpsychol Kinderpsychiatr. 2019 Jan;68(1):27-42. doi: 10.13109/prkk.2019.68.1.27. German. PMID 30628875